CLINICAL TRIAL: NCT01706471
Title: Safety and Efficacy of the Early Introduction of Everolimus (Certican®) With Low Dose of Cyclosporine in de Novo Kidney Recipients After 1 Month of Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2009-0109
Record Dates: First submitted 2012-10-08; First posted 2012-10-15 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Planned Kidney Transplantation
Keywords: verLowCNI
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everolimus + Low dose CsA +PD (Experimental)
  Interventions: Drug: Everolimus + Low dose CsA +PD
- Myfortic+ Standard CsA + PD (Active Comparator)
  Interventions: Drug: Myfortic+ Standard CsA + PD

INTERVENTIONS:
Drug: Everolimus + Low dose CsA +PD — Group A : Initiation of 5mg/kg bid Neoral dose and 720mg bid Myfortic and then adjusting Neoral targeting 150-200ng. After 1 month reduce Neoral dose as following table and Certican starting 0.75mg bid then adjust Certican 3-8ng/ml. Myfortic continue until Certican trough level goes up >3 ng/mL. Steroid dose follows local protocol.
  Arms: Everolimus + Low dose CsA +PD
Drug: Myfortic+ Standard CsA + PD — Group B : Initiation of 5mg/kg bid Neoral dose and 720mg bid Myfortic and then adjusting Neoral targeting 150-200ng/ml. After 1 month reduce Neoral dose targeting 100-200ng with no change of Myfortic dose. Steroid dose follows local protocol.
  Arms: Myfortic+ Standard CsA + PD

SUMMARY:
Calcineurin inhibitors, such as cyclosporine and tacrolimus, have improved allograft survival in kidney organ transplantation. Indeed, they have reduced the incidence of acute rejection episodes of cadaveric allograft recipients. Although marked progression has been made in initial survival rates, long-term kidney graft survival has yet to show such encouraging results. Because CNIs are associated with adverse effects, particularly nephrotoxicity, which contribute to declining organ function and eventual graft loss. In kidney transplants, progressive allograft dysfunction has been shown to develop in as many as 94% of patients by 1 year.

Therefore, reducing or eliminating the dose of CNIs to minimize nephrotoxicity must be balanced against the maintenance of adequate immunosuppression.

Certican allows CNI dose reduction then provides renal function improvement and current PSI strategy point out that early intervention is important in managing the risk of CAN before it develops in both de novo and maintenance renal transplant recipients.

To demonstrate Certican early introduction after 1 month provides better renal function with no change of efficacy compared to standard regimen, and also prevent delayed wound healing.

ELIGIBILITY:
Inclusion Criteria:

1. Males or Females aged 18~65 years
2. De novo recipients of cadaveric, living unrelated or living related donor kidney transplants
3. Received kidney transplant from aged 10~65years donor
4. Willing to provide written informed consent
5. Completing study visits according to study protocol

Exclusion Criteria:

1. Recipients of multiple organ transplants
2. Kidney transplant from non-heart beating cadaveric donor / organ donor after cardiac death
3. Recipients of A-B-O incompatible transplants or lymphocyte cross-match positive transplants
4. Recipients of extra-renal solid organ transplants or stem cell transplants
5. Recipient/ donor who are known to have anti-HCV, HIV or HBsAg positive
6. Diagnosed as Cancer within the past 5 years (except complete recovered squamous cell or basal cell skin cancer)
7. Drug Hypersensitivity to investigational drugs or related drugs Females are pregnant and lactating
8. Any of the following laboratory abnormalities at screening:

   * ALT, AST, ALP, total bilirubin > 3 times the upper limit
   * ANC < 1,500mm3 or WBC < 2,500mm3 or platelet < 100,000 mm3
   * Cholesterol > 350 mg/dl or 9.0 mmol/L, TG > 500 mg/dl or 5.6mmol/L

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Reduced Exposure Cyclosporine in Renal Transplant Recipients | 12 months after the time of kidney transplantation
  A 12-month, multi center, randomized, open-label, non-inferiority study of efficacy and safety comparing early introduction of Certican® after 1 month and standard regimen in de novo renal transplant recipients

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Yonsei University College of Medicine, Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Oh CK, Huh KH, Ha J, Kim YH, Kim YL, Kim YS. Safety and efficacy of the early introduction of everolimus with reduced-exposure cyclosporine a in de novo kidney recipients. Transplantation. 2015 Jan;99(1):180-6. doi: 10.1097/TP.0000000000000225. PMID 24983307